CLINICAL TRIAL: NCT01002066
Title: Rapid Malaria Diagnostic Tests in Fever Patients Attending Primary Health Care Facilities in Zanzibar - Effectiveness as Diagnostic and Surveillance Tool in the New Context of Low Malaria Endemicity
Brief Title: Effectiveness Of Rapid Diagnostic Tests in the New Context of Low Malaria Endemicity in Zanzibar
Acronym: RDTACT
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Zanzibar Malaria Control Programme (Other Government); World Health Organization (Other)
Responsible Party: Principal Investigator, Anders Björkman, Professor, Karolinska University Hospital
Other Study IDs: ACT2010
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2011-11

CONDITIONS: Fever; Malaria
Keywords: Fever; Malaria; RDT; IMCI; Children<5 years of age; ACT
MeSH Terms: conditions — Fever; Malaria

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Whole blood collected on Rapid diagnostic tests (RDT)s and Filter paper (FP)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to study the effectiveness of wide scale RDT use at the primary health care level in previously high malaria endemic area during malaria pre-elimination phase for improved targeting of anti-malarial drugs, malaria surveillance and epidemic alertness.

DETAILED DESCRIPTION:
During the last 6 years Zanzibar has undergone a dramatic change in malaria epidemiology and burden of disease, with a marked decline of Plasmodium falciparum malaria among febrile children from approximately 30% to 1% or below and a reduction of crude child mortality of 50% Overuse of the expensive ACTs will not only be a substantial financial burden on the health care system in Zanzibar, but will also spur anti-malarial drug resistance with devastating effect on global malaria control efforts and prevent other causes of fever from being appropriately treated, e.g. pneumonias which require antibiotics. Rapid Diagnostic Tests (RDTs), based on antigen detection of P. falciparum, are proposed as a future cornerstone to improve diagnostic efficiency also at the peripheral health care level beyond the reach of microscopy services

IMCI algorithms based on clinical symptoms could potentially be made more efficient and cost effective if simple parasitological diagnostic methodologies were incorporated. Zanzibar is among the first regions to incorporate RDT in the IMCI guidelines in Africa, which provides a unique research opportunity to scientifically evaluate the effectiveness of incorporating RDT in the existing IMCI algorithm.

Another key challenge for Zanzibar is to monitor potential development of parasite resistance to ACT when the number of malaria positive patients is insufficient to conduct standard in vivo efficacy trials. We propose that RDT could play a critical new role also in this regard.

ELIGIBILITY:
Inclusion Criteria:

* All patients >2 months of age with confirmed fever, with a measured axillary temperature of ≥37.5˚C, or history of fever within the preceding 24 hours
* Presenting to the health facility from 8.00 to 16.00 Monday to Friday.
* Informed consent

Exclusion Criteria:

* Previous enrolment in the study within the last 28 days.
* Severe disease that requires immediate referral as defined by the clinician

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary health care units (PHCUs) and Primary health care centres (PHCCs) in North A and Micheweni Districts in Zanzibar
Sampling Method: Non-Probability Sample
Enrollment: 3890 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Adherence to Rapid diagnostic tests (RDT) result | Five months

CONTACTS AND LOCATIONS:
Overall Officials: Anders Björkman, Professor, Principal Investigator — Karolinska University Hopsital; Andreas Mårtensson, Ph.D, M.D., Principal Investigator — Karolinska University Hospital; Kristina Elfving, M.D., Principal Investigator — Karolinska University Hospital; Mwinyi Msellem, MSc, Principal Investigator — Zanzibar Malaria Control Programme; Delér Shakely, M.D., Principal Investigator — Karolinska University Hopsital
Locations (1):
- Primary health care centers (PHCC)s and Primary health care units (PHCUs), Kivunge and Micheweni, Zanzibar, Tanzania

REFERENCES:
- [Derived] Shakely D, Elfving K, Aydin-Schmidt B, Msellem MI, Morris U, Omar R, Weiping X, Petzold M, Greenhouse B, Baltzell KA, Ali AS, Bjorkman A, Martensson A. The usefulness of rapid diagnostic tests in the new context of low malaria transmission in Zanzibar. PLoS One. 2013 Sep 4;8(9):e72912. doi: 10.1371/journal.pone.0072912. eCollection 2013. PMID 24023791